CLINICAL TRIAL: NCT05918289
Title: Effectiveness of Blended Active Aging Education Program on Active Aging Factors and Wellbeing in Community-dwelling Older Adults in Pakistan. A Randomized Control Trail
Brief Title: Improving Wellbeing in Older Adults: The Impact of an Active Aging Education Program in Pakistan
Acronym: BAAEP
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhengzhou University (Other)
Responsible Party: Principal Investigator, Rashida Bibi, Principal Investigator, Zhengzhou University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 52
Record Dates: First submitted 2023-05-10; First posted 2023-06-26 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: Aging Well; Well Aging; Quality of Life; Well-Being, Psychological
Keywords: Active aging; education program; older adults; Pakistan
MeSH Terms: conditions — Psychological Well-Being

STUDY DESIGN:
Intervention Model Description: This model is focusing on active aging through didactic including information on active aging and aging well, positive thinking, mindful eating, reflection on life, physical exercises, practical group activities, video-guided exercises, a booklet for a home for practice
Masking Description: The trainers were unknown of the data collection and results, they are unaware of the research objective, and research hypothesis.
  The data collectors are unaware of the purpose of the study and the intention to treat the mechanism, data analyzer is unaware of the outcome of the results and unaware of which coding number for which group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention and control (Experimental): Treatment group taken intervention of education program designed for elders and the control group did not take any intervention but at the end of the time duration they were taken the opportunity of 3 days class room intervention
  Interventions: Behavioral: Blended& integrated happy aging active aging program(BIHAAAP)

INTERVENTIONS:
Behavioral: Blended& integrated happy aging active aging program(BIHAAAP) — 12 Weeks intervention devided in to two phases( face to face and home based)

SUMMARY:
The goal of this randomized control trial study is to evaluate the effect of the happy aging education program on active aging determinants, and quality of life among community-based Muslim older adults compared with the control group who avail only health education.

Q1.• What is the effect of the BIHAAAP on physical, mental, and behavioral aspects of active aging among community-dwelling older adults in the compression to the control group who only avail health education? Q2. What is the effect of the BAAEP on the quality of life among community-dwelling older adults in Pakistan?

Treatment: (1) Face-to-face: 6 days, (2) home-based 12 weeks.

1. Face to Face: (1) Orientation, the aging process, the importance of exercises in old age, coping strategies, and the beneficial effects of body movements in Muslim prayers. (2) Hands-on training regarding proper body movement in Muslim five-time prayers.
2. Home-based treatment: (1) A Pictorial booklet consisting of tips to spend happy life in old age and a workbook to complete. (2) Audio video recorded by a physiotherapist on the proper body movements in five-time prayers to follow at home shared through whats app number of at least one family member if the person does not have a smartphone.

Comparison group: One-day orientation. After the trial, the control group availed of the booklet and video-recorded Muslim prayers-like exercises.

DETAILED DESCRIPTION:
Road Map of the Study Development of BAAEP Development of content for face-to-face training consisted of lectures, group activities, and hand on practice with the intention to improve physical, mental, cognitive, and behavioral approaches for active aging.

Booklet contents: Tips on mindfulness eating habit practice to mentally prepare for any food items before eating, positive thought generation practice by different scenarios, benefits of exercises in pictorial form, pictures of healthy couples and beneficial effects of relationships, tips for spiritual health, and the booklet contents homework after each session.

Video development Detail about Muslim prayers like exercises

* Prepared guidelines from two published papers along with comprehensive descriptions regarding each picture to develop a video on the mimic Muslim prayer's body movements' video for home practice.
* Appointment of a physiotherapist holding a Masters's degree and practicing as a physiotherapist in a private rehabilitation center, the checklist was shared to practice.
* The physiotherapist will develop an outline to develop a video and will arrange a meeting with other two physiotherapists, one doctor, and one community health nurse. The major focus was to assess any restrictions for elders with any disease. The physiotherapist will develop a video by adding instructions in the local language.
* A series of movements consisting of body parts movement starting from deep two deep breaths.
* Movement of neck, shoulders, hands and arms, head, feet, and every joint of the body. It will take only 10 to 15 minutes. The structured exercise steps follow all the steps mentioned in the traditional Islamic prayers and yoga breathing. The detail of the Muslim Salat-like exercise is mentioned below
* 1: Standing and Takbir: Takbir, is the movement of raising hands to the level of one's face so that the thumbs touch the ear lobule, by doing that taking one deep breath, precedes another prayer posture.
* 2: The Standing (Qiyam): Fundamental standing position for up to 60-90 seconds, with some exceptions such as wrapping the arms in front of the belly in such a way that the scapula is slightly retracted, taking two deep breaths. The chin is tucked in and the person looks at his feet while standing, resulting in flexion at the upper cervical spine, thus activation of the deep neck flexors, which are prone to getting weak as in upper cross syndrome[50].
* 3: Rukuk: The bowing, or Rukuk, is a very important position biomechanically in which forward bending occurs at the thoracic and lumbar spines, which leads to the stretching of the Para spinal muscles and structures. The trunk and the lower extremity are at an approximately 90-degree angle to each other. The person attempts to look between his toes while adopting this position, which results in the activation of deep neck flexors, which are usually prone to getting weak. The hip joint is in flexion, the knees are extended, and the ankle is at 90° with the lower leg as in standing. The shoulders are slightly flexed and the elbows are fully extended, whereas the hands rest on the knees. The average duration of a Rukuk may last up to 10-15 seconds along
* 4: Prostration ( Sajdah): The prostration posture of Salat is similar to a fetus's pose, and flexion occurs at the thoracic and lumbar spines, accompanied by hip flexion. The knees are in mid-flexion, the ankle is in the neutral position, and the toes are extended. The shoulders are slightly abducted, the elbows in mid-flexion, and the wrists extended with the palms parallel to the ears. The lower cervical spine is also slightly extended during prostration. It strengthen the triceps brachii and showed the greatest activation. Triceps brachial activation in Salah was also significantly higher than in the child's pose.
* The Sitting (Tahiyyat/Jalsa) Posture of Salat: The sitting (taqiyya) two-time head position involves sitting on the floor with the lumbar and thoracic spines in neutral, the hip joint in flexion, and the knee joint in full flexion for up to 30-60 seconds. This results in a stretching of the quadriceps Femoris muscle. The hands are placed on the distal aspect of the anterior thigh, with shoulders flexed and elbows extended, though the full extension is not present, along with slight extension at the wrists.
* Turning of head side by side: Cervical exercises. Turns the head to both shoulders fit right and then left.

Study Area: Study setting: Two residential areas of Peshawar, Khyber Pakhtunkhwa

1. Sample selection process: Lady health workers (LHWs) will be approached through the District health office Peshawar and identified households with elders aged> 60 years from the family registration registers of each LHW.Identified 300 older adults in the jurisdiction of haji camp, skandertown, and Tarnab form.

   Conduct a general health awareness program for all elders who registered with the five LHWs and will be given the responsibility of monitoring elders to perform exercises in their homes. A convenient sampling method will be used to recruit some of the elderly in the two regions of Peshawar in Khyber Pakhtunkhwa province.
2. Recruitment of the participant 2.1. Sample size calculation: Sample size will be calculated using G-power by priori power analysis. An effect size of 0.83 will be used from a previous study conducted on technology-based elder education. The sample size calculation will assume (i.e. α =0.05, power=0.8. Total 140.

   2.2. Screening for eligibility: We will conduct a health awareness program in three high schools at different times in which around 300 elders participated. Arranged three points in which all elders were checked for cognitive, activity, auditory, and visual impairment levels.

   2.2.1. Preliminary screening: screening will be conducted by physiotherapists and community health nurses for frailty, and severe health problems for example cardiac problems, cognitive problems auditory and severe visual problems (referred to psychologist, ENT specialist, and family medicines doctor.

   2.2.2 Secondary screening: To register for trial the screening will be taken to take ( consent, registration, baseline assessment for sedentary lifestyles who reported spending less than 20 to 30 minutes per week outside in their home in the past month.

   2.3. Sampling technique= Computer generated sequence will be employed to randomize study subjects either to intervention or control group and then a web-based data management system using a permuted block algorithm (with random block lengths) stratified by sex.

   2.4. Treatment group=70, Control group=70 2.5. Treatment group= BAAEP, C= Usual activities Participants included: (a) sedentary retired adults aged 65 and older who reported spending less than 20 min per week in the past month
3. Procedure for implementation of treatment/ intervention 3.1. face: Three trainers(physiotherapist, community health nurse, psychologist) conducted the face-to-face sessions after getting training and piolet study. A PowerPoint presentation was prepared according to the protocol. piloting was done in the same setting to modify the discrepancies after taking feedback.

The setting was checked for ventilation, temperature, lighting, and chairs. 3.1.1. Setting for intervention: Three government high schools and one private high school were allocated for the training sessions by taking approval from the district education officer and the honor of a private school.

3.1.2. Three volunteers will be assigned for the setting and technical support through proper agreement. The generator was arranged for power backup during the session.

3.13.3. Interventions process: Orientation and three sections (1) didactic such as giving information and knowledge regarding aging, challenges and positive aspects of aging),(2) group activity for positive thinking, joke as an energizer, discussion on hobbies and interest,(3) hands-on training for( mind fullness and prayers like proper body movements exercises. Each group consisted of 15 participants, five-session in a day and each group availed 90 minutes sessions per week.

During the session continue feedback will be taken from the participants regarding any difficulty in performing exercises, understanding level, and further suggestions.

3.13.Transforming from face-to-face sessions to home-based training

* Make a list of the WhatsApp numbers of each participant
* Research group will share the videos one by one with their numbers
* Booklets will be distributed and take signatures and kept records for both video and booklet distribution.
* Lady heath visitors along with the research team will be responsible to make sure of the implementation at home and recording any adverse effects. Reporting and referring forms were developed and given to the research team for recording.

Quality control: Homogeneous population characteristics; both male and female; data collectors and data analysts will be kept unaware of the research intention.

Participants were not blind due to the ethical considerations of the study. Researchers were not directly involved in the session and only observed the ongoing process, the researchers were not involved in the data collection process only randomly checking the objectivity, and researchers were not directly involved in data analysis to prevent biases. A person who will be unaware of the purpose of the study performed randomization of the total 140 elders in two groups. The research team was not aware of the outcome variables and was not involved in the data collection task. The data collectors were kept blind from the intervention strategies.

The study protocol is approved by the School of Nursing, Zhengzhou University. Written approval was taken from the School of Nursing, ZZU, and from the local health department of Khyber Pakhtunkhwa. Approval was taken from the local government of the province along with the readiness of the research teams and area representatives for conducting the session inside their premises of the area.

All participants were informed about the study and a written approval of willingness was taken from all the participants. In addition, their personal details are kept secret by assigning ID numbers and did not be used for any other purposes and this was well ensured.

ELIGIBILITY:
Inclusion Criteria:• Both males and females aged 60 or above

* Independent Older adults
* No visual and auditory impairments
* Local people who understand the local language(Urdu)
* No serious conditions
* Physically and mentally fit
* Availability of digital resources( smartphone, computer or Television) to play video at home
* Healthy volunteers

Exclusion Criteria:• Dependent older adults

* Visual and Auditory Impairments
* Non-local people who are unable to understand the local language
* Serious Conditions
* Physically and mentally impaired
* Unwillingness to participate

Ages: 60 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 140 (Actual)
Dates: Start 2022-08-15 (Actual); Primary Completion 2022-11-15 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Active aging level | 12 weeks
  The active aging scale will be used to assess the overall active aging, consisting of self-reliance, healthy lifestyle, social contribution, participation in leisure activities, developing spiritual wisdom, strengthening family ties, and a sense of economic security. The scale consisted of 29 items with seven factors, using the 5 Likert scale 1-5 scoring method, where the total score range is 29 to 128 points. A score <64 indicates poor aging, 64 to 96 points indicates that the level of active aging is moderate, and a higher score of 96 indicates a higher level of active aging.
Sense of well-being | 12 Weeks
  One commonly used tool to measure the sense of well-being was developed by the World Health Organization( WHO-5 Well-Being Index), consisting of five items that assess positive mood, vitality, and general well-being. Each item is rated on a 5-point Likert scale, ranging from 0 (not present) to 5 (constantly present). The scores <15 consider poor well-being, 15 to 20 Mild well-being problems, and > 20 scores will be regarded as high well-being.
Time Up and Go test. | 12 weeks
  Time Up and Go test scores: scores were assigned to go and back sit down for which 10 to 19 seconds were considered normal, 20 to 29 in the gray list included in fall risk, and >30 dependent considered high risk for fall.
  .
Physcial functional ability test | 12 weeks
  Berg balance test. Berg balance scale scoring ranges from 0 to 56. The lower your score, the more at risk of losing balance. Scoring method;0 to 20: A person with a score in this range will likely need the assistance of a wheelchair to move around safely; 21 to 40: A person with a score in this range will need some type of walking assistance, such as a cane or a walker; 41 to 56: A person with a score in this range is considered independent

CONTACTS AND LOCATIONS:
Locations (1):
- Zhengzhou University, Zhengzhou, Henan, China

IPD SHARING:
Plan to Share IPD: No